CLINICAL TRIAL: NCT06971731
Title: A Phase 3, Double-Blind, Randomized, Two-Period, Multicenter, Placebo-Controlled, Efficacy and Safety Study of JNT-517 for the Treatment of Participants With Phenylketonuria
Brief Title: A Study to Evaluate the Safety and Efficacy of JNT-517 in Participants With Phenylketonuria (PKU)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JNT517-301
Record Dates: First submitted 2025-05-07; First posted 2025-05-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Drug: JNT-517 - 150 mg BID (Tablet) (Experimental)
  Interventions: Drug: JNT-517 Tablet
- Drug: JNT-517 - 75 mg BID (Tablet) (Experimental)
  Interventions: Drug: JNT-517 Tablet
- Placebo - BID (Placebo Comparator): One-third (1/3) of participants in the study will be assigned to placebo BID during Treatment Period Part 1. After 6 weeks, these participants will transition to Treatment Period Part 2 and receive JNT-517 at 150 mg BID for 46 weeks.
  Interventions: Drug: Placebo Tablet: BID

INTERVENTIONS:
Drug: JNT-517 Tablet — JNT-517: 75 mg BID
  Arms: Drug: JNT-517 - 75 mg BID (Tablet)
Drug: JNT-517 Tablet — JNT-517: 150 mg BID
  Arms: Drug: JNT-517 - 150 mg BID (Tablet)
Drug: Placebo Tablet: BID — Placebo Tablet: BID
  Arms: Placebo - BID

SUMMARY:
The goal of this Phase 3, randomized study is to assess the safety, efficacy, tolerability, and pharmacokinetics (PK) of oral JNT-517 in adults (18 years of age or older) with PKU. Participants will receive either JNT-517 or placebo and will be blinded to their treatment assignment. Participants will have a 2 in 3 (or approximately 67%) chance of receiving JNT-517 during the first part of the study which will last approximately six weeks. During the second part of the study every participant who continues in the study will receive one of two doses of JNT-517 for an additional 46 weeks. The study requires a screening period of up to 35 days to ensure dietary stabilization and amino acid levels required to meet study eligibility. In total, participation in the study could last for up to 400 days.

Participants will:

Take 75 mg JNT-517 or 150 mg JNT-517, or a placebo BID (2x per day) for approximately 365 days; Visit the clinic or have a mobile health nurse visit your home for checkups and tests; Collect urine sample at home and bring to clinic on specified days; Keep a food diary 3 days before each study visit

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥18 years of age on Day 1
2. Clinical diagnosis of PKU
3. Average of at least 3 plasma Phe levels (after >4-hour fast) during Screening period of ≥360 μmol/L
4. Not on pegvaliase within 4 weeks prior to Screening
5. If on sapropterin or large neutral amino acids, such as PheBloc®, NeoPhe®, and PreKunil® at Screening, must be on a stable dose 4 weeks prior to Screening and for the entire study duration.
6. Willing and able to maintain a stable diet in Phe and total protein (intact protein and medical food protein) and able to adjust diet through the duration of the study according to the Dietary Management Guidelines
7. Body weight >45 kg
8. If biologically female of childbearing potential:

   1. Must have a negative serum pregnancy test at Screening and a negative urine pregnancy test by Day 1
   2. Must practice sexual abstinence, or if involved in any sexual intercourse that could lead to pregnancy, must agree to use 2 highly effective contraceptive methods from Screening until at least 30 days after the last study drug administration
   3. If taking estrogen- or progesterone-based oral contraceptives, must agree to use 2 other highly effective methods of contraception or must agree to sexual abstinence during the study
   4. Must refrain from donating ova during the course of the study and for 30 days after the last dose of the study drug.
9. If a biologically female not of childbearing potential or postmenopausal, defined as follows:

   1. Has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy)
   2. Has had amenorrhea for minimum of 1 year with confirmation by levels of follicle stimulating hormone testing
   3. Has not achieved menarche (has not had first menstrual period). If a female achieves menarche during the study, she will need to follow the contraception requirement for females of childbearing potential
10. If biologically male, must practice sexual abstinence, or if involved in any sexual intercourse that could lead to pregnancy, must agree to use highly effective contraceptive methods from Day 1 until at least 30 days after the last study drug administration and must refrain from donating sperm during the course of the study and for 30 days after the last dose of the study drug NOTE: No restrictions are required for biological males who have undergone a documented vasectomy at least 4 months prior to Screening. If the vasectomy procedure is not documented or was performed less than 4 months prior to Screening, males must follow the same contraception as for non-vasectomized participants.
11. Participants with psychiatric illness must be well-controlled for the last 6 months prior to the Screening visit and if on medication, on stable medications for the last 3 months.
12. Capable of giving signed informed consent or parent/legal guardian to provide informed consent and the participant to give assent and confirm able to comply with study procedures

Exclusion Criteria:

* Exclusion Criteria

Participants will be excluded from the study if any of the following criteria are met:

1. Any acute or uncontrolled chronic medical condition that would prevent the participant from complying with the procedures or place the participant at risk if they participate in the study
2. Positive for hepatitis B or C or human immunodeficiency virus
3. Any history of malignancy of any organ system (other than non-melanoma skin cancer or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases
4. Any history of significant liver disease
5. Any history of cataracts or more than minimal cataracts observed during the Screening ophthalmologic examination. Minimal cataracts are defined as changes similar to lens opacities classification system III (LOCS III), lens grade C1, N1 or P1
6. Any surgical or medical conditions that may affect study drug absorption, distribution, metabolism, or excretion
7. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 by 2021 Chronic Kidney Disease Epidemiology Collaboration formula
8. Participation in another investigational drug trial within 30 days or, if known, 5 half-lives of the investigational drug (whichever is longer). For gene therapy or editing trials, participants must have received the intervention >6 months prior to Screening visit and with stable plasma Phe in the past 2 months prior to Screening visit.
9. Alcohol consumption within 5 days of randomization and/or unwilling to limit to 1 alcoholic drink per day until after the 6-month study visit
10. History of drug/alcohol abuse in the last year
11. Use of any medications that are inhibitors or inducers of cytochrome P450 (CYP3A4) or inhibitors of the transporter P-glycoprotein (P-gp) within 4 weeks prior to randomization and unwilling and/or unable to avoid these medications throughout the treatment duration (Appendix A)
12. Use of any medications that are substrates of breast cancer resistance protein (BCRP), multidrug and toxin extrusion (MATE)1, or MATE2-K within 4 weeks prior to randomization and unwilling and/or unable to avoid these medications throughout the treatment duration (Appendix A) NOTE: Participants will be permitted to continue with estrogen- or progesterone-based oral contraceptives, but must agree to use 2 other methods of contraception, where at least 1 must be highly effective, or must agree to sexual abstinence during the study.
13. Current, recent, or suspected active viral or bacterial infection within 2 weeks prior to and during the Screening Period
14. Unable to tolerate oral medication or have a condition that would interfere with the absorption of JNT-517
15. Allergy to JNT-517 or any component of the investigational product
16. Any of the following laboratory values at the Screening visit: -Alanine aminotransferase or aspartate aminotransferase values >1.5× the upper limit of normal (ULN)-Total bilirubin ˃ULN unless history of Gilbert Syndrome and then total bilirubin >4 mg/dL is exclusionary-Hemoglobin <11.0 g/dL (<110.0 g/L)-White blood cell count >ULN-Platelets <150 × 109/L (<150,000/mm3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Percent change in plasma phenylalanine (Phe) levels from baseline to mean of Weeks 2, 4, and 6 in the JNT-517 150 mg BID dose group | Baseline visit to Week 6

SECONDARY OUTCOMES:
Participants achieving plasma Phe <600 μmol/L at end of Period 1 among those with baseline ≥600 μmol/L in the 150 mg BID and 75 mg BID groups, respectively | Baseline visit to Week 6
Participants achieving plasma Phe levels <360 μmol/L at end of Period 1 in the 150 mg BID and 75 mg BID groups, respectively | Baseline visit to Week 6
Percent change in plasma Phe from baseline to mean of Weeks 2, 4, and 6 of Period 1 in the JNT-517 75 mg BID group | Baseline visit to Week 6
Participants achieving plasma Phe levels <120 μmol/L at end of Period 1 in the JNT-517 75 mg BID and 150 mg BID dose groups, respectively | Baseline visit to Week 6
Change in plasma Phe from baseline to Weeks 2, 4, and 6 of Period 1 in the JNT-517 75 mg BID and 150 mg BID dose group, respectively | Baseline visit to Week 6

CONTACTS AND LOCATIONS:
Locations (15):
- United States (6):
  - University of Florida (UF) Health Shands Hospital, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health (UTHealth) Science Center at Houston, Houston, Texas
  - Utah Health - The University of Utah Hospital, Salt Lake City, Utah
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Mater Health - Mater Hospital Brisbane, South Brisbane
- Centre Hospitalier Régional Universitaire (CHRU) de Tours - Hôpital Bretonneau, Tours, France
- Japan (2):
  - Nihon University Hospital, Chiyoda-ku
  - Osaka Metropolitan University Hospital, Osaka
- Netherlands (2):
  - Universitair Medisch Centra (AMC)- Amsterdam, Amsterdam
  - Beatrix Children's Hospital, Groningen
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com